CLINICAL TRIAL: NCT03831009
Title: Weight-bearing Radiographs to Evaluate Stability in Ankles With Isolated Trans-syndesmotic Lateral Malleolar (Weber Type B) Fractures. A Pilot Study.
Brief Title: Weight-bearing Radiographs to Evaluate Stability in Ankles With Isolated Weber Type B Fractures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18/07031-7; 2018/1585/REK sør-øst B (Other Grant/Funding Number: Regional Committees for Medical and Health Research Ethics)
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-06

CONDITIONS: Lateral Malleolus Fractures; Ankle Fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment. Based on stability evaluation using weight-bearing adiographs one group recieves surgery, one group recieves non-surgical treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Weight-bearing stable/Gravity stable (Active Comparator): Ankles that are considered stable using weight-bearing radiographs AND gravity stress test will be assigned to conservative treatment
  Interventions: Other: Conservative treatment
- Weight-bearing stable/Gravity unstable (Active Comparator): Ankles that are considered stable using weight-bearing radiographs but unstable using gravity stress test will be assigned to conservative treatment
  Interventions: Other: Conservative treatment
- Weight-bearing unstable/Gravity unstable (Active Comparator): Ankles that are considered unstable using weight-bearing radiographs AND gravity stress test will be assigned to open reduction internal fixation (ORIF)
  Interventions: Procedure: Open reduction internal fixation (ORIF)
- Weight-bearing unstable/Gravity stable (Active Comparator): Ankles that are considered unstable using weight-bearing radiographs but stable using gravity stress test will be assigned to open reduction internal fixation (ORIF)
  Interventions: Procedure: Open reduction internal fixation (ORIF)

INTERVENTIONS:
Procedure: Open reduction internal fixation (ORIF) — Open fracture reduction followed by internal fixation using a plate and screws. The goal is an osteosynthesis that allow for early range-of-motion exercises, but weightbearing is usually not tolerated until 6 weeks postoperatively.
  Arms: Weight-bearing unstable/Gravity stable; Weight-bearing unstable/Gravity unstable
Other: Conservative treatment — Conservative treatment involves ankle protection with a functional brace (AirCast) for 6 weeks. Participants will be instructed to bear weight as tolerated and to actively do standardized range-of-motion exercises.
  Arms: Weight-bearing stable/Gravity stable; Weight-bearing stable/Gravity unstable

SUMMARY:
The investigators will conduct a prospective cohort study on the use of weight-bearing radiographs to evaluate stability in ankles with isolated, trans-syndesmotic (Weber type B) fibular fractures. Stable fractures will be treated conservatively using a functional brace, unstable fractures will undergo surgical fixation.

DETAILED DESCRIPTION:
It is widely accepted that fractures in stable ankles can be treated non-operatively and fractures in unstable ankles needs internal fixation surgery (Michelson, Magid & McHale, 2007, Gougoulias, Khanna, Seellariou, Maffulli, 2010). Clinical decision-making is thus based on ankle stability evaluation. The integrity of medial structures, mainly the deep deltoid ligament, is considered the most important determinant for stability of the ankle mortise (Michelson, Magid & McHale, 2007, Gougoulias, Khanna, Seellariou, Maffulli, 2010). Weber B fractures, with no obvious sign of medial side injury on initial plain radiographs, have to be considered of uncertain stability until adequate stress testing is performed.

Currently there is no definite consensus on what test(s) best determines stability in ankles with undisplaced, isolated lateral malleolar fractures. Much used methods comprises manual stress radiographs and gravity stress radiographs (McConnel, Creevy & Tornetta, 2004). However recent studies have shown that such methods overestimate the need for surgical fixation indicating the need for a different method to make up the basis for surgical indication (Dawe, Shafafy, Quayle, Gougoulias, Wee & Sakellariou, 2015, Hastie, Akhtar, Butt, Baumann & Barrie, 2015, Holmes, Acker, Murphy, McKinney, Kadakia & Irwin, 2016, Hoshino, Nomoto, Norheim & Harris, 2012, Koval, Egol, Cheung, Goodwin & Spratt (2007), Seidel et al., 2017, Weber, Burmeister, Flueckiger & Krause, 2010). Authors of recent studies have proposed weightbearing radiographs as an alternative method to distinguish stable and unstable fractures, significantly reducing the need for operative treatment (Dawe et al., 2015, Hastie et al., 2015, Hoshino et al, 2012, Holmes et al., 2016, Seidel et al., 2017, Weber et al. 2010).

To evaluate weight-bearing radiographs ability to determine stability our primary focus is to evaluate if conservative treatment for "gravity unstable/weightbearing stable" ankles produces different outcomes than conservative treatment for "gravity stable/weightbearing stable" ankles.

Participants will be assigned to non-operative or surgical treatment based on ankle stability evaluation using results from weightbearing radiographs consistently. Stable ankles will be treated non-operatively with a functional brace (AirCast) for 6 weeks. Participants will be instructed to bear weight as tolerated and to actively do standardized range-of-motion exercises. Standard operative treatment is open reduction and internal fixation of the fracture using plate and screws.

ELIGIBILITY:
Inclusion Criteria:

* Isolated Weber type B fractures without radiological signs of medial clear space widening on initial radiographs. Patients must be 18-80 years of age. Before the injury patients should be mobilized without walking aids. They should be compliant with good communication skills in the Norwegian or English languages. Patients must live in Østfold or nearby areas so they are able to meet to follow-up consultations.

Exclusion Criteria:

* Patients presenting with any of the following will be excluded from the study: Fracture of the medial malleolus. Information about prehospital fracture closed reduction. Open fracture. Fracture resulting from high-energy trauma or multi-trauma. Pathologic fracture. Diabetes Mellitus type 1 and 2. Neuropathies. Cognitive disorders. Previous history of ankle fracture. Previous history of ankle-/foot surgery. Generalized joint disease such as RA. Patients with insufficient Norwegian or English language proficiency or lack of communication skills.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The Manchester-Oxford Foot Questionnaire (MOxFQ) | 24 months
  Ankle/foot specific patient-reported outcome measure

SECONDARY OUTCOMES:
Olerud-Molander Ankle Score (OMAS) | 24 months
  Ankle/foot specific patient-reported outcome measure. Maximum score (100) = best. Minimum score = 0 (worst). Poor = 0-30, Fair = 31-60, Good = 61-90, Excellent = 91-100. Presented as total score (0-100).
AOFAS ankle-hindfoot | 24 months
  Ankle/foot specific patient-reported outcome measure
VAS/NRS of pain | 24 months
  Visual analogue pain scale - patient reported. Scale 0-10. 10 = worst possible pain, 0 = no pain
Eq-5d | 24 months
  Genereic health related quality of life patient reported outcome measure
Fracture healing | 24 months
  Radiographic result
Registration of complications | 24 months
  Yes/No for malalignment, deep vein trobosis, nerve injury, wound infection, delayed wound healing and crossover to surgery (including reason for crossover).
Bilateral ankle range-of-motion | 24 months
  Measured in degrees with a goniometer ad modum Lindsjö.
Bilateral calf circumference | 24 months
  Calf circumference in centimeters measured 10 cm distal to the tibial tubercle Calf circumference in centimeters measured 10 cm distal to the tibial tubercle using measuring tape

CONTACTS AND LOCATIONS:
Overall Officials: Marius Molund, Principal Investigator — Ostfold Hospital Trust
Locations (1):
- Østfold Hospital Trust, Sarpsborg, Østfold fylke, Norway

REFERENCES:
- See also: REC study registration — https://helseforskning.etikkom.no/prosjekterirek/prosjektregister/prosjekt?p_document_id=1062903&p_parent_id=1067266&_ikbLanguageCode=n